CLINICAL TRIAL: NCT05591976
Title: The Effects of Exercise Training on Fitness, Function and Quality of Life in Youth With Inflammatory Bowel Disease: A Pilot Study
Brief Title: Exercise Training in Youth With Inflammatory Bowel Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Brian Timmons, Professor, McMaster University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 13-194
Record Dates: First submitted 2022-09-20; First posted 2022-10-24 (Actual); Last update posted 2022-10-24 (Actual); Status verified 2022-10

CONDITIONS: Pediatric Inflammatory Bowel Diseases; Pediatric Crohns Disease; Pediatric Ulcerative Colitis
MeSH Terms: conditions — Pediatric ulcerative colitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise group (Experimental): Participants are assessed for outcomes prior to intervention, mid-way through intervention and immediately after intervention.
  Interventions: Other: Exercise training program

INTERVENTIONS:
Other: Exercise training program — 16-week, structured exercise training program including resistance and aerobic exercise

SUMMARY:
Children and adolescents with inflammatory bowel disease (IBD) suffer from many extra-intestinal side effects, including impaired muscle strength, low aerobic fitness, low bone density, and chronic inflammation. While exercise training can help remedy these issues in adults with IBD, no studies have examined the physiological effects of a structured aerobic and resistance exercise training intervention for youth with IBD.

The aim of this pilot study is to to assess the feasibility, safety, and participant satisfaction of a structured 16-week training program for children with IBD. The secondary objectives of this study were to quantify the effects of a 16-week exercise training program on select physiological and behavioural outcomes in children with IBD.

ELIGIBILITY:
Inclusion Criteria:

* In remission (score of >10) according to the pediatric Crohn's disease activity index (PCDAI) or the ulcerative colitis activity index (PUCAI)
* Confirmed IBD diagnosis

Exclusion Criteria:

* Children who exercise train 3 times a week of more

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 11 (Actual)
Dates: Start 2013-05-01 (Actual); Primary Completion 2014-06-01 (Actual); Study Completion 2014-06-01 (Actual)

PRIMARY OUTCOMES:
Recruitment | Change from baseline at 8 weeks and 1 week post intervention
  Measure of patient recruitment (number of patients approached, enrolled, refused)
Retention | Change from baseline at 8 weeks and 1 week post intervention
  Percent of patients that completed the study after enrolment
Adherence | Change from baseline at 8 weeks and 1 week post intervention
  Percent of prescribed exercise completed across sessions
Compliance | Change from baseline at 8 weeks and 1 week post intervention
  Percent of exercise sessions completed
Changes in IBD-related symptoms: Pediatric Ulcerative Colitis Activity Index | Change from baseline at 8 weeks and 1 week post intervention
  Tracking changes in IBD-related symptoms based on Pediatric Ulcerative Colitis Activity Index (scored 0-85, where higher score indicates more severe disease)
Changes in IBD-related symptoms: Pediatric Crohn's Disease Activity Index | Change from baseline at 8 weeks and 1 week post intervention
  Tracking changes in IBD-related symptoms based on Pediatric Crohn's Disease Activity Index (scored 0-100, where higher score indicates more severe disease)
Qualitative assessment of participant likes and dislikes of the training program and suggestions for improvement | Change from baseline at 8 weeks and 1 week post intervention
  Assessed by qualitative interview looking at likes and dislikes of the training program as well as suggestions for improvement
Tracking adverse events | During training session
  Adverse events are event that occurs during the course of exercise training that cause the participant physical or psychological harm

SECONDARY OUTCOMES:
Body mass composition absolute values | Change from baseline at 8 weeks and 1 week post intervention
  Lean body mass (kg), fat body mass (kg), bone mineral content (kg), total mass (kg) all measured by Dual X-ray Absorptiometry scan
Body mass composition as a percent of total body mass | Change from baseline at 8 weeks and 1 week post intervention
  Lean body mass (% of total mass), fat body mass (% of total mass), bone mineral content (% of total mass). Absolute body composition measures (kg) divided by total body mass (kg) make % of total mass. All measured by Dual X-ray Absorptiometry scan.
Bone mineral density | Change from baseline at 8 weeks and 1 week post intervention
  Bone mineral density (g/cm^3) measured by Dual X-ray Absorptiometry scan.
Aerobic fitness: maximum rate of oxygen consumption attainable during physical exertion | Change from baseline at 8 weeks and 1 week post intervention
  VO2 peak (L*min-1) measured by the McMaster All-Out Progressive Continuous Cycling Test using a calibrated metabolic cart
Aerobic fitness: peak workload | Change from baseline at 8 weeks and 1 week post intervention
  peak workload (watts) measured by the McMaster All-Out Progressive Continuous Cycling Test using a cycle ergometer
Aerobic fitness: peak heart rate | Change from baseline at 8 weeks and 1 week post intervention
  Peak heart rate (beats*min-1), measured by the McMaster All-Out Progressive Continuous Cycling Test using heart rate monitor
Muscle strength | Change from baseline at 8 weeks and 1 week post intervention
  Grip strength (Nm), isokinetic and isometric leg strength (Nm) and isokinetic and isometric arm strength (Nm) all measured with an isokinetic dynamometer
Physical activity levels | Change from baseline at 8 weeks and 1 week post intervention
  Time spent in physical activity (at light, moderate and high intensity) and sedentary time (min*day-1) measured by a waist-worn accelerometer
Inflammatory cytokine levels | Change from baseline at 8 weeks and 1 week post intervention
  IL-6 and TNF-alpha concentrations (pg/ml) measured from patient plasma by enzyme-linked immunosorbent assays

CONTACTS AND LOCATIONS:
Overall Officials: Brian Timmons, PhD, Principal Investigator — McMaster University
Locations (1):
- McMaster Children's Hospital, Hamilton, Ontario, Canada